CLINICAL TRIAL: NCT06539741
Title: Mechanisms of Variability in the Analgesic Response to Ibuprofen Following Third Molar Extraction
Brief Title: Variability in Analgesic Response to Ibuprofen
Status: Recruiting | Type: Observational
Sponsor: University of Pennsylvania (Other)
Collaborators: National Institute of Dental and Craniofacial Research (NIDCR) (NIH)
Responsible Party: Sponsor
Other Study IDs: 856367; 1R01DE033405-01A1 (NIH)
Record Dates: First submitted 2024-08-01; First posted 2024-08-06 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Impacted Third Molar Tooth; Pain, Acute
MeSH Terms: conditions — Acute Pain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Plasma, serum, urine, whole blood, peripheral blood mononuclear cells, stool, oral microbiome, tissue
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Complete Responders: Patients who do not require supplemental opioids, in addition to a standard-of-care NSAID-based pain management regimen, for pain relief following third molar extraction
- Partial Responders: Patients who require supplemental opioids (oxycodone 5 mg), in addition to a standard-of-care NSAID-based pain management regimen, for pain relief following third molar extraction

SUMMARY:
Nonsteroidal anti-inflammatory drugs (NSAIDs), like ibuprofen, are recommended as first-line treatment for post-surgical dental pain. However, there is variability in analgesic response, and some patients require supplemental opioids for adequate pain relief. The goal of this study is to identify the factors that contribute to the need for opioid after third molar extraction to help limit unnecessary opioid prescriptions in patients who will have good pain relief with ibuprofen alone.

DETAILED DESCRIPTION:
The dramatic increase in opioid prescriptions over the past years has been linked to the concomitant rise in opioid addiction and to deaths from opioid abuse. Young adults' initial exposure to opioid analgesics is often following extraction of their impacted third molars, with an average of 5,000,000 cases in the USA per year. Over-prescribing of opioids for surgical pain, often 2-5 times more than patients actually use, further exacerbates this problem, as patients tend to save leftover pills rather than discard them. Up to 70% of individuals who become addicted to prescription opioids had access to leftover pills prescribed for others. This is particularly troubling as the odds of transitioning to heroin from prescription opioid abuse are much higher than other suspected gateway drugs, about 40 fold greater than non-gateway drug users.

Multiple studies have demonstrated that non-addicting nonsteroidal anti-inflammatory drugs (NSAIDs) such as ibuprofen and diclofenac are effective in relieving pain after dental impaction surgery, being at least equally efficacious as optimal doses of immediate release opioid formulations combined with acetaminophen. However, these assessments of pain relief represent average scores and approximately 22% and 50% of individuals required additional opioid-containing rescue analgesics when ibuprofen and diclofenac were employed at FDA-approved dosages. A deeper understanding of the sources of variability in pain relief should allow improvements in the overall efficacy of NSAIDs by targeting treatment to those who are most likely to receive sufficient pain relief. Thus, optimizing pain therapy with NSAIDs by personalization would be expected to help limit the unnecessary prescription of highly addicting immediate release opioids. Moreover, these results may have applicability to other types of pain that are driven by inflammation.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated informed consent form
2. Stated willingness to comply with all study procedures and availability for the duration of the study
3. Ability to take oral medication and be willing to adhere to the study treatment regimen
4. Men and women greater than 18 years of age requiring extraction of at least one impacted mandibular third molar tooth (at least 50% covered with bone).
5. Absence of other major medical problems or contraindications to surgery or study drugs.
6. Female subjects of child bearing potential must be using a medically acceptable method of contraception (oral contraception, Depo-Provera injection, IUD, condom with spermicide, diaphragm, cervical cap, progestin implant, abstinence, tubal ligation, oophorectomy, TAH) throughout the entire study period. All female subjects must consent to a urine pregnancy test at screening and a urine pregnancy test on the day of surgery, which must be negative at all time points.
7. Has not ingested caffeine-containing products within 12 hours of surgery.
8. All subjects must consent to a urine drug test at screening. Results must be negative (except for THC) unless the subject is on a stable dose of a non-analgesic drug for a legitimate medical purpose. A positive test for THC will be permitted and the frequency of use will be documented. A positive result will be reported to the subject.
9. Does not consume more than 1 alcoholic beverage per day on average.
10. Subjects must reach a level of at least moderate pain within four hours of surgery completion, with a pain score greater than or equal to 4 on a 0-10 numerical pain scale
11. Subjects must be willing and able to complete safety and efficacy diaries.
12. An escort must be available to pick up the subject at the end of at the end of the surgical/dosing visit (Visit #2).

Exclusion Criteria:

1. Female subjects who are pregnant or nursing a child.
2. Subjects who have received an investigational drug or used an experimental medical device within 30 days prior to screening, or who gave a blood donation of ≥ one pint within 8 weeks prior to screening.
3. Subjects who are sensitive or allergic to ibuprofen, acetaminophen, or their components.
4. Subjects who are sensitive or allergic to aspirin or other NSAIDs.
5. Subjects who are sensitive or allergic to oxycodone or other opioids (excluding nausea and constipation).
6. Presence of a serious medical condition (e.g. poorly controlled hypertension or diabetes, gastrointestinal disorders such as bleeding ulcer, coagulation or bleeding disorders, significantly impaired cardiac, renal, hepatic, respiratory, or thyroid function) that according to the investigator may interfere with interpretation of the study results or compromise the safety of a potential subject.
7. Acute local infection at the time of surgery that could confound post-surgical evaluation.
8. Use of any confounding prescription or non-prescription drug within 24 hours of the surgical procedure, including analgesics, sedating antihistamine, sedative, alcohol, or CNS/psychotropic agents (i.e. sleep aids, benzodiazepines). Hormonal contraceptives, hormone replacement therapy (including males taking testosterone as a hormone replacement to treat a documented low testosterone level), or thyroid replacement hormones are allowed. Individuals taking other/additional chronic stable medications can be considered on a case-by-case basis for inclusion in the study if agreed upon by judgment of the investigator.
9. Subjects with any abnormal laboratory value or physical finding that according to the investigator may interfere with interpretation of the study results, be indicative of an underlying disease state, or compromise the safety of a potential subject.
10. Subjects who have a history of opioid use disorder or other substance use disorder, based upon history and judgment of the Investigator.
11. Subjects who are unwilling to provide a blood sample for genetic analyses.
12. Employees of the principal investigator, sub-investigators, or relative of an employee who is directly involved in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients presenting for surgical extraction of partial or full bony impacted mandibular third molars at the Oral Surgery Clinics at Penn Dental Medicine
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-01-03 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Supplemental Opioid Use | Up to 7 days after third molar extraction
  Use of oxycodone in addition to ibuprofen + acetaminophen

SECONDARY OUTCOMES:
Gene Expression Profiling | Up to 7 days after third molar extraction
  mRNA levels will be measured in peripheral blood mononuclear cells
COX-1 activity | Up to 7 days after third molar extraction
  COX-1 activity will be measured ex vivo using a whole blood assay and in vivo by quantifying concentrations of prostaglandin metabolites in urine.
COX-2 activity | Up to 7 days after third molar extraction
  COX-2 activity will be measured ex vivo using a whole blood assay and in vivo by quantifying concentrations of prostaglandin metabolites in urine.
DNA sequencing | 1 day
  Assessment of genetic variation
Pain intensity score | Up to 7 days after third molar extraction
  Rating of pain from 0 (no pain) to 10 (worst imaginable pain)
Inflammatory mediator profiling | Up to 7 days after third molar extraction
  Assessment of cytokines in plasma
Complete blood count with differential | Up to 7 days after third molar extraction
  Assessment of proportions of red blood cells, white blood cells, and platelets in whole blood

CONTACTS AND LOCATIONS:
Overall Officials: Katherine N Theken, PharmD, PhD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania School of Dental Medicine, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No